CLINICAL TRIAL: NCT02027025
Title: Study of SPARC1103 in Subjects With Spasticity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_11_03
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Spasticity
Keywords: Spasticity, Multiple sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPARC 1103 low dose (Active Comparator): The subjects will receive SPARC 1103 low dose
  Interventions: Drug: SPARC1103 low dose
- SPARC1103 high dose (Active Comparator): The subjects will receive SPARC1103 high dose
  Interventions: Drug: SPARC1103 high dose
- SPARC Placebo (Placebo Comparator): The subjects will receive SPARC Placebo
  Interventions: Drug: SPARC Placebo

INTERVENTIONS:
Drug: SPARC1103 low dose — once daily
  Arms: SPARC 1103 low dose
Drug: SPARC1103 high dose — once daily
  Arms: SPARC1103 high dose
Drug: SPARC Placebo
  Arms: SPARC Placebo

SUMMARY:
Study of SPARC1103 in subjects with spasticity

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than or equal to 18 years of age
* Willing to sign the informed consent form
* Women of child bearing potential willing to practice an acceptable method of birth control
* Known history of spasticity due to MS

Exclusion Criteria:

* Administration of an investigational drug or device within 30 days prior to Screening Visit 1
* Unable to comply with trial procedures in the opinion of the Investigator
* Concomitant neurologic conditions causing spasticity
* Any medical condition, including psychiatric disease or epilepsy, which would interfere with the interpretation of the trial results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (15):
  - SPARC Site 4, Long Beach, California
  - SPARC Site 6, San Diego, California
  - SPARC Site 10, Aurora, Colorado
  - SPARC Site 2, Jacksonville, Florida
  - SPARC Site 15, Miami, Florida
  - SPARC Site 7, Miami Springs, Florida
  - SPARC Site 5, Orlando, Florida
  - SPARC Site 13, Tampa, Florida
  - SPARC Site 11, Kansas City, Kansas
  - SPARC Site 3, Lenexa, Kansas
  - SPARC Site 1, Bingham Farms, Michigan
  - SPARC Site 14, Albuquerque, New Mexico
  - SPARC Site 9, Charlotte, North Carolina
  - SPARC Site 8, Cleveland, Ohio
  - SPARC Site 12, Richland, Washington
- Russia (5):
  - SPARC Site 18, Moscow
  - SPARC Site 17, Nizhny Novgorod
  - SPARC Site 20, Samara
  - SPARC Site 19, Smolensk
  - SPARC Site 16, Ufa
- Ukraine (3):
  - SPARC Site 22, Dnipro
  - SPARC Site 21, Ivano-Frankivsk
  - SPARC Site 23, Lviv

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- SPARC1103 Low Dose: SPARC1103 low dose dosing regimen:
  1 capsule orally, approximately 30 minutes
- SPARC1103 High Dose: SPARC1103 high dose dosing regimen
  1 capsule orally, approximately 30 minutes
- SPARC Placebo: SPARC Placebo dosing regimen
  1 capsule orally, approximately 30 minutes
Period: Overall Study
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo
Started | 48 | 47 | 47
Completed | 47 | 42 | 46
Not Completed | 1 | 5 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Sponsor's decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SPARC1103 Low Dose: Age: 50.5 (9.12)
- SPARC1103 High Dose: Age: 52.3 (9.33)
- SPARC Placebo: Age: 50.2 (10.43)
- Total: Total of all reporting groups
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo | Total
Number analyzed (Participants) | 48 | 47 | 47 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (9.12) | 52.3 (9.33) | 50.2 (10.43) | 51.0 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 28 | 80
  Male | 25 | 18 | 19 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 2 | 5 | 16
  White | 37 | 45 | 42 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 47 | 47 | 142

OUTCOME MEASURES:

1. Primary Outcome: Least Square Mean Difference (Placebo Versus Each SPARC1103 Dose) in Change From Baseline in Modified Ashworth Score
Description: The modified Ashworth scale is a 6-point scale as follows:
  Minimum score of 0 (better outcome) = no increase in tone Maximum score of 4 (worst outcome) = affected part(s) rigid in flexion or extension
  For calculation of modified Ashworth Score, the following scores were assigned to each category of modified Ashworth scale: not testable=NA, 0=0 units, 1=1 unit, 1+ = 2 units, 2 = 3 units, and 4 = 5 units. The total score was the sum of the scores of the 6 lower extremity muscle groups on both left and right sides (range = o0 to 60).
Time Frame: Baseline, Day 24
Population: Intent to treat population: SPARC1103 low dose, N=47; SPARC 1103 high hose, N=42; and Placebo, N=46
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- SPARC1103 Low Dose: Least square mean difference (Placebo versus SPARC 1103 low dose) in change from baseline in total modified Ashworth score on day 24
- SPARC1103 High Dose: Least square mean difference (Placebo versus SPARC 1103 high dose) in change from baseline in total modified Ashworth score on day 24
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose
Number analyzed (Participants) | 47 | 42
score on a scale | 0.33 (1.47) | 0.03 (1.53)

2. Secondary Outcome: Least Square Mean Difference (Placebo Versus Each SPARC1103 Dose) in Change From Baseline in Night Time Awakening Score
Description: Nighttime awakening score was assessed as follows:
  The subject was asked the following question on the morning of Day 24: How many times did you wake up last night due to spasticity? Score range from "0" (better score) to "infinity" (worse score)
Time Frame: Baseline, Day 24
Population: Intent to treat population: SPARC 1103 low dose, N=47; SPARC 1103 high dose, N=42; and Placebo N=46.
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Groups:
- SPARC1103 Low Dose: Least square mean difference (Placebo versus SPARC 1103 low dose) in change from baseline in nighttime awakening score on day 24
- SPARC1103 High Dose: Least square mean difference (Placebo versus SPARC 1103 high dose) in change from baseline in nighttime awakening score on day 24
- SPARC Placebo: Change from baseline for nighttime awakening score on day 24
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo
Number analyzed (Participants) | 47 | 42 | 46
Awakenings | -0.25 (0.449) | -0.24 (0.470) | 0.23 (0.449)
Statistical Analysis 1: Comparison: SPARC1103 Low Dose vs SPARC Placebo; Test type: Superiority; p = 0.4532, ANCOVA; LS mean difference = -0.48, 95% CI 2-sided [-1.73 to 0.78], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: SPARC1103 High Dose vs SPARC Placebo; Test type: Superiority; p = 0.4704, ANCOVA; LS mean difference = -0.47, 95% CI 2-sided [-1.76 to 0.82], Standard Error of Mean 0.65

3. Secondary Outcome: Least Square Mean Difference (Placebo Versus Each SPARC1103 Dose) in Change From Baseline in Spasm Frequency
Description: Spasm frequency was assessed using following 4-point scale as follows:
  Minimum score of 0 (better outcome))=no spasm Maximum score of 4 (worst outcome)=Spasms occurring more than 10 times per hour
Time Frame: Baseline, Day 24
Population: Intent to treat population:
  SPARC 1103 low dose, N= 47; SPARC1103 High dose, N=42; and Placebo, N=46
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- SPARC1103 Low Dose: Least square mean difference (Placebo versus SPARC 1103 low dose) in change from baseline in spasm frequency on day 24
- SPARC1103 High Dose: Least square mean difference (Placebo versus SPARC 1103 high dose) in change from baseline in spasm frequency on day 24
- SPARC Placebo: Least square mean change from baseline in spasm frequency on day 24
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo
Number analyzed (Participants) | 47 | 42 | 46
score on a scale | -0.46 (0.129) | -0.46 (0.140) | -2.6 (0.133)
Statistical Analysis 1: Comparison: SPARC1103 Low Dose vs SPARC Placebo; Test type: Superiority; p = 0.3013, ANCOVA; LS mean difference = -0.19, 95% CI 2-sided [-0.56 to 0.17], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: SPARC1103 High Dose vs SPARC Placebo; Test type: Superiority; p = 0.2994, ANCOVA; LS mean difference = -0.20, 95% CI 2-sided [-0.58 to 0.18], Standard Error of Mean 0.19

4. Secondary Outcome: Clinical Global Impression of Change Results at 24 Hours Post Dose on Day 24
Description: The clinician (other than the one performing the Modified Ashworth Scale assessment) rated his/her overall (global) impression of change in spasticity using the 7-point scale shown below:
  Minimum score of 1 (better outcome) = very much improved Maximum score of 7 (very much worse) = very much worse
Time Frame: Baseline, Day 24
Population: Intent to treat population:
  SPARC 1103 low dose, N=47; SPARC 1103 high dose, N=42; and Placebo N=46
Measure: Number; unit: participants
Groups:
- SPARC1103 Low Dose; SPARC1103 High Dose; SPARC Placebo: Clinical global impression of change results at 24 hours post dose on Day 24
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo
Number analyzed (Participants) | 47 | 42 | 46
participants
  CGIC - very much improved | 4 | 2 | 3
  CGIC - much improved | 12 | 8 | 8
  CGIC - minimally improved | 16 | 20 | 26
  CGIC - no change | 11 | 6 | 7
  CGIC - minimally worse | 3 | 5 | 2
  CGIC - much worse | 1 | 1 | 0
  CGIC - very much worse | 0 | 0 | 0
Statistical Analysis 1: Comparison: SPARC1103 Low Dose vs SPARC Placebo; Test type: Superiority; p = 0.3815, Chi-squared
Statistical Analysis 2: Comparison: SPARC1103 High Dose vs SPARC Placebo; Test type: Superiority; p = 0.7491, Chi-squared

5. Secondary Outcome: Subject Global Impression of Severity of Spasticity
Description: The subject was asked "Overall, how would you rate the severity of your spasticity over the past 24 hours?"
  The 7-point scale for Subject's global impression of severity assessment is as follows:
  minimum score of 1 = normal, no spasticity maximum score of 7 (worst outcome)= worst spasticity imaginable
Time Frame: Baseline, Day 24
Population: Intent to treat population: SPARC1103 low dose, N=47; SPARC1103 high dose, N=42; and Placebo, N=46
Measure: Count of Participants; unit: Participants
Groups:
- SPARC1103 Low Dose; SPARC1103 High Dose; SPARC Placebo: Subject's global impression of severity of spasticity at Day 24
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo
Number analyzed (Participants) | 47 | 42 | 46
Participants
  Normal - no spasticity | 5 | 4 | 4
  Borderline spasticity | 4 | 5 | 6
  Mild spasticity | 15 | 19 | 15
  Moderate spasticity | 19 | 12 | 18
  Marked spasticity | 4 | 1 | 2
  Severe spasticity | 0 | 1 | 1
  Worst spasticity imaginable | 0 | 0 | 0
Statistical Analysis 1: Comparison: SPARC1103 Low Dose vs SPARC Placebo; Test type: Superiority; p = 0.8991, Chi-squared
Statistical Analysis 2: Comparison: SPARC1103 High Dose vs SPARC Placebo; Test type: Superiority; p = 0.8829, Chi-squared

ADVERSE EVENTS:
Time Frame: Screening through Day 24
Groups:
- SPARC1103 Low Dose; SPARC1103 High Dose; SPARC Placebo: Subjects with treatment emergent adverse events
Arm/Group | SPARC1103 Low Dose | SPARC1103 High Dose | SPARC Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/47 | 0/47
Other Adverse Events (participants affected / at risk) | 4/48 | 2/47 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC1103 Low Dose (N=48) | SPARC1103 High Dose (N=47) | SPARC Placebo (N=47)
Influenza (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC1103 Low Dose (N=48) | SPARC1103 High Dose (N=47) | SPARC Placebo (N=47)
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
headache (Nervous system disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT02027025/Prot_SAP_000.pdf